CLINICAL TRIAL: NCT01788176
Title: Phase 2 Study - The Use of a Single 5 mg Dose of Zoledronic Acid in Complex Regional Pain Syndrome Patient.
Brief Title: The Use of Zoledronic Acid to Complex Regional Pain Syndrome
Acronym: Aclasta
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Pérola Grinberg Plapler, MD, PhD, Director of Physical Medicine Division Of Institute Orthopedics and Traumatology of University of Sao Paulo General Hospital, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446HBR10T
Record Dates: First submitted 2012-10-09; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Complex Regional Pain Syndromes; drug therapy; zoledronic acid
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): One single intravenous infusion of 100ml of saline (placebo control group).
  Interventions: Drug: Placebo
- Zoledronic acid (Active Comparator): one single dose of 5mg intravenous infusion of zoledronic acid (interventional group)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — One single dose of 5mg intravenous infusion of zoledronic acid (interventional group)
  Arms: Zoledronic acid
Drug: Placebo — one single intravenous infusion of 100ml of saline.
  Arms: Saline

SUMMARY:
To evaluate the efficacy and the safety of using a single, intravenous 5mg dose of zoledronic acid in managing pain in Complex Regional Pain Syndrome patients.

DETAILED DESCRIPTION:
Complex regional pain syndrome (CRPS) is a disorder of the extremities that is characterized by spontaneous unexplained disproportionate pain, hyperalgesia, swelling, limited range of motion, vasomotor instability, skin changes, and patchy bone demineralization.The incidence of CRPS was estimated to be 5.46 per 100,000 person years at risk in Olmsted County, Minnesota (US), with a prevalence of 20.57 per 100,000, while its incidence in the general population of the Netherlands was estimated to be much higher, at 26.2 per 100,000 person-years. The adverse effects were not serious and lasted just a few days. The beneficial effects of other bisphosphonates have been already documented in several placebo-controlled trials; however, there are no reports on the use of zoledronic acid to reduce pain in CRPS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age of both genders, with continuing pain that is disproportionate to any inciting event, with cardinal features of CRPS.
2. Pain - after initial injury with signs and symptoms present at first visit
3. History of previous unsuccessful treatment for pain, with a minimum of two drug therapies, such as non steroidal anti-inflammatory drugs, steroids, antidepressants, central acting analgesics, calcitonin or sympathetic blocks, (not bisphosphonates) for at least six months.
4. Must report at least one symptom in three of the four following categories:

   1. Sensory: Reports of hyperesthesia and/or allodynia
   2. Vasomotor: Reports of temperature asymmetry and/or skin color changes and/or skin color asymmetry
   3. Sudomotor/Edema: Reports of edema and/or sweating changes and/or sweating asymmetry
   4. Motor/Trophic: Reports of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin).
5. Must display at least one sign* at time of evaluation in two or more of the following categories:

   1. Sensory: Evidence of hyperalgesia (to pinprick) and/or allodynia (to light touch and/or deep somatic pressure and/or joint movement)
   2. Vasomotor: Evidence of temperature asymmetry and/or skin color changes and/or asymmetry
   3. Sudomotor/Edema: Evidence of edema and/or sweating changes and/or sweating asymmetry
   4. Motor/Trophic: Evidence of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin).
6. Skin temperature of the affected side equal or higher than on the non-affected side.
7. No other diagnosis better explains the signs and symptoms.

Exclusion Criteria:

1. Presence of systemic diseases including diabetes mellitus, hyperthyroidism, renal and liver dysfunction, peripheral vascular or cardiovascular diseases, uncontrolled hypertension, rheumatoid and hematopoietic diseases, neurological diseases not related to CRPS, overt alcohol addiction, positive pregnancy test and/or lactating women, hyperparathyroidism, and hypocalcaemia.
2. Creatinine clearance <35mL/min, with serum creatinine measured before the dose of zoledronic acid.
3. Pre-existing hypocalcaemia and disturbance of mineral metabolism (e.g. hyperparathyroidism, thyroid surgery, parathyroid surgery, malabsorption syndromes, and excision of small intestine).
4. Hypersensitivity to zoledronic acid or any component drugs used in the trial.
5. Patients with asthma and aspirin-sensitivity
6. Pregnancy or unwillingness to use contraceptive methods during the trial
7. Patients who have previously used any kind of bisphosphonate, especially zoledronic acid.
8. Osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain measured on Visual Analog Scale | up to 12 months after treatment

SECONDARY OUTCOMES:
Lower Limbs vertical force on Wii platform | Baseline, 3, 6 and 12 months
American Orthopaedic Foot and Ankle Scale (AOFAS) | Baseline, 3, 6 and 12 months after treatment
36-Item Short Form Health Survey (SF-36) | Baseline, 3, 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linamara R. Battistella, PHD, Study Director — Centro de Pesquisa Clínica do Instituto de Medicina Física e de Reabilitação do Hospital das Clínicas da FMUSP
Locations (1):
- Centro de Pesquisa Clínica do Instituto de Medicina e Reabilitação do HCFMUSP, São Paulo, São Paulo, Brazil